CLINICAL TRIAL: NCT00934895
Title: Phase I/II Study of Weekly Abraxane and RAD001 in Women With Locally Advanced or Metastatic Breast Cancer. A Study of the Cancer Institute of New Jersey Oncology Group (CINJOG)
Brief Title: Phase I/II Study of Weekly Abraxane and RAD001 in Women With Locally Adv. or Metastatic Breast Ca
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed early due to slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Toppmeyer, MD, Professor, CINJ, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro0220090058; P30CA072720 (NIH); CDR0000648116 (Other: NIH); Pro0220090058 (Other: IRB); CRAD001C2448; (Other: Novartis); NCI-2012-00547 (Other: CTRP (Clinical Trials Reporting Program)); 040803 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Results first posted 2022-11-07 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; HER2-negative breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase I / Phase II (Experimental): Phase I:
  * Abraxane will be given by IV for 30 minutes on the first day of the first three weeks of each 28 day cycle.
  * RAD001 will be given by tablet. The first group of patients will receive RAD001 once daily depending on side effects seen drug could be increased later to twice a day for a 28 day cycle.
  Once a safe and effective drug range is established, the study moves into Phase II.
  Phase II:
  The maximum tolerated dose (established in Phase I) will be given as scheduled below and we will measure the effectiveness of the study drug combination.
  * Abraxane will be given by IV (intravenous infusion) for 30 minutes on the first day of the first three weeks of each 28 day cycle (Day 1, Day 8, and Day 15 of each cycle).
  * RAD001 will be given by tablet based on the dose established in the Phase I part of the study.
  Interventions: Drug: everolimus; Drug: abraxane

INTERVENTIONS:
Drug: everolimus — Orally administered RAD001 will be initiated at 5 mg daily. Each cohort Phase I: administration will proceed based on escalation criteria. RAD001 will be given initially once every day. Doses will be adjusted per the dosing regimen for each cohort throughout the Phase I portion of the study
  Other Names: RAD001
Drug: abraxane — Doses of Abraxane will be calculated on Day 1 of each cycle using the patient's actual weight in the determination of body surface area. A variance of 5% of the calculated total dose will be allowed.
  Other Names: nab paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving paclitaxel albumin-stabilized nanoparticle formulation together with everolimus may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of everolimus when given together with paclitaxel albumin-stabilized nanoparticle formulation and to see how well it works in treating women with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose and recommended phase II dose of everolimus when administered in combination with paclitaxel albumin-stabilized nanoparticle formulation in women with locally advanced or metastatic breast cancer. (Phase I)
* To determine the antitumor activity of this regimen, as measured by clinical tumor response according to RECIST criteria, in these patients. (Phase II)

Secondary

* To determine the safety and tolerability of everolimus when administered at the recommended phase II dose in combination with paclitaxel albumin-stabilized nanoparticle formulation in these patients.

OUTLINE: This is a multicenter, phase I dose-escalation study of everolimus followed by a phase II study.

Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Patients also receive oral everolimus once daily or once every other day on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Locally recurrent or metastatic disease
  * Not amenable to surgery or radiotherapy
* HER2/neu-negative disease
* Has ≥ 1 measurable lesion, as defined by RECIST criteria

  * No non-measurable lesions (e.g., pleural effusion or ascites) other than bone metastases

    * Bone metastases as the sole site of disease allowed provided there are ≥ 2 lytic bone lesions by x-ray, CT scan, or MRI
  * Lesions irradiated in the advanced setting are not considered sites of measurable disease unless clear tumor progression has been documented in these lesions since the completion of radiotherapy
* No bilateral diffuse lymphangitis carcinomatosa of the lung (> 50% of lung involvement) or evidence of liver metastases estimated as involving > one third of the liver by sonogram and/or CT scan
* No unstable CNS metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin > 9 g/dL
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (≤ 5 times ULN in patients with liver metastases)
* INR < 1.5 times ULN
* Serum creatinine ≤ 1.5 mg/dL
* Fasting serum cholesterol ≤ 300 mg/dL (or 7.75 mmol/L) (levels outside this threshold allowed provided statin therapy is initiated)
* Fasting triglycerides ≤ 2.5 times ULN (levels outside this threshold allowed provided statin therapy is initiated)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

  * Oral, implantable, or injectable contraceptives are not considered effective contraception
* No ascites or encephalopathy due to liver disease
* No neuropathy ≥ grade 2
* No impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of everolimus, including any of the following:

  * Ulcerative disease
  * Uncontrolled nausea, vomiting, or diarrhea
  * Malabsorption syndrome
* No active, bleeding diathesis
* No known HIV seropositivity
* No known hypersensitivity to everolimus or sirolimus (rapamycin), paclitaxel albumin-stabilized nanoparticle formulation, or lactose
* No history of noncompliance to medical regimens
* No severe and/or uncontrolled medical condition or other condition that could affect study participation, including any of the following:

  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within the past 6 months, or serious uncontrolled cardiac arrhythmia
  * Severely impaired lung function
  * Active (acute or chronic) or uncontrolled infections or disorders
  * Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by study treatment
  * Liver disease (e.g., cirrhosis, chronic active hepatitis, or chronic persistent hepatitis)
* No other malignancies within the past 5 years, except curatively treated carcinoma in situ of the cervix or nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

* Prior systemic endocrine therapy for advanced breast cancer allowed
* No prior chemotherapy for advanced breast cancer

  * Prior adjuvant chemotherapy allowed
* No prior small bowel resection
* More than 5 days since prior strong CYP3A inhibitors or inducers (e.g., rifabutin, rifampin, clarithromycin, ketoconazole, itraconazole, voriconazole, ritonavir, or telithromycin)
* More than 30 days since prior radiotherapy and recovered (alopecia allowed)
* Prior localized radiotherapy for analgesic purposes allowed provided radiotherapy has been completed and the patient's condition is stabilized
* No prior radiotherapy to ≥ 25% of the bone marrow
* More than 30 days since prior investigational drugs
* More than 1 week since prior and no concurrent immunization with attenuated live vaccines
* No concurrent oral anti-vitamin K medication, except low-dose coumadin
* No concurrent systemic steroids or other immunosuppressive agents as chronic therapy

  * Topical applications, inhaled sprays, eye drops, or local injections allowed
  * A short duration (< 2 weeks) of systemic corticosteroids allowed
* No concurrent hormone replacement therapy, topical estrogens (including any intra-vaginal preparations), megestrol acetate, or selective estrogen-receptor modulators (e.g., raloxifene)
* No other concurrent investigational or anticancer agents
* Concurrent antiangiogenic agents allowed
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-07-15 (Actual); Primary Completion 2014-01-07 (Actual); Study Completion 2015-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L. Toppmeyer, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (3):
- United States (3):
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Rutgers Cancer Institute of New Jersey (Hamilton), Hamilton, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey Oncology Group. They study was open to accrual on 07/15/2009 and closed to accrual on 01/07/2014.
Pre-assignment Details: We are reporting results on 27 eligible patients. One patient was deemed ineligible.
Groups:
- Phase I Level -1 - RAD001 5mg Daily, Abraxane 60mg/m2: Phase I:
  * Abraxane 60 mg/m2 will be given by IV for 30 minutes on the first day of the first three weeks of each 28 day cycle.
  * RAD001 will be given by tablet (5 mg). The first group of patients will receive RAD001every day depending on side effects seen drug could be increased later to twice a day for a 28 day cycle.
  Once a safe and effective drug range is established, the study moves into Phase II.
- Phase 1 Level -2 - RAD001 5mg Every Other Day, Abraxane 60mg/m2: Phase I:
  * Abraxane 60 mg/m2 will be given by IV for 30 minutes on the first day of the first three weeks of each 28 day cycle.
  * RAD001 will be given by tablet (5 mg). The first group of patients will receive RAD001every other day depending on side effects seen drug could be increased later to twice a day for a 28 day cycle.
  Once a safe and effective drug range is established, the study moves into Phase II.
- Phase 1 Level 0 RAD001 5mg Daily, Abraxane 80mg/m2: Phase I:
  * Abraxane 80 mg/m2 will be given by IV for 30 minutes on the first day of the first three weeks of each 28 day cycle.
  * RAD001 will be given by tablet (5 mg). The first group of patients will receive RAD001 every day depending on side effects seen drug could be increased later to twice a day for a 28 day cycle.
  Once a safe and effective drug range is established, the study moves into Phase II.
- Phase 1 Level 1 RAD001 5mg Daily, Abraxane 100mg/m2: Phase I:
  * Abraxane 100 mg/m2 will be given by IV for 30 minutes on the first day of the first three weeks of each 28 day cycle.
  * RAD001 will be given by tablet (5 mg). The first group of patients will receive RAD001 every day depending on side effects seen drug could be increased later to twice a day for a 28 day cycle.
  Once a safe and effective drug range is established, the study moves into Phase II.
- Phase 1 Level 2 RAD001 5mg Daily, Abraxane 125mg/m2: Phase I:
  * Abraxane 125 mg/m2 will be given by IV for 30 minutes on the first day of the first three weeks of each 28 day cycle.
  * RAD001 will be given by tablet (5 mg). The first group of patients will receive RAD001 every day depending on side effects seen drug could be increased later to twice a day for a 28 day cycle.
  Once a safe and effective drug range is established, the study moves into Phase II.
- Phase 1 Level 3 RAD001 10mg Daily, Abraxane 125mg/m2: Phase I:
  * Abraxane 125 mg/m2 will be given by IV for 30 minutes on the first day of the first three weeks of each 28 day cycle.
  * RAD001 will be given by tablet (10 mg) daily. The first group of patients will receive RAD001 every day depending on side effects seen drug could be increased later to twice a day for a 28 day cycle.
  Once a safe and effective drug range is established, the study moves into Phase II.
- Phase II Abraxane at 150 mg/m2: The Phase II treatment schedule will continue following the same 28 day cycle schedule as Phase I.
  Abraxane will be administered without premedication as a 30 minute intravenous infusion weekly for the first 3 of the 4 weeks of a 28 day cycle (Day 1, Day 8, and Day 15 of each cycle). The dose of Abraxane to be used in the Phase II portion of the trial will be based upon the MTD established in the Phase I portion of this trial.
  RAD001 will be administered on the schedule and at the maximum tolerated dose as determined by the Phase I results.
Period: Overall Study
Arm/Group | Phase I Level -1 - RAD001 5mg Daily, Abraxane 60mg/m2 | Phase 1 Level -2 - RAD001 5mg Every Other Day, Abraxane 60mg/m2 | Phase 1 Level 0 RAD001 5mg Daily, Abraxane 80mg/m2 | Phase 1 Level 1 RAD001 5mg Daily, Abraxane 100mg/m2 | Phase 1 Level 2 RAD001 5mg Daily, Abraxane 125mg/m2 | Phase 1 Level 3 RAD001 10mg Daily, Abraxane 125mg/m2 | Phase II Abraxane at 150 mg/m2
Started | 0 | 0 | 3 | 6 | 4 | 0 | 14
Completed | 0 | 0 | 3 | 6 | 4 | 0 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: no data available to analyze.
Groups:
- Phase II: Phase II:
  The maximum tolerated dose (established in Phase I) will be given as scheduled below and we will measure the effectiveness of the study drug combination.
  * Abraxane will be given by IV (intravenous infusion) for 30 minutes on the first day of the first three weeks of each 28 day cycle (Day 1, Day 8, and Day 15 of each cycle).
  * RAD001 will be given by tablet based on the dose established in the Phase I part of the study.
  everolimus: Orally administered RAD001 will be initiated at 5 mg daily. Each cohort Phase I: administration will proceed based on escalation criteria. RAD001
- Total: Total of all reporting groups
Arm/Group | Phase I Level -1 - RAD001 5mg Daily, Abraxane 60mg/m2 | Phase 1 Level -2 - RAD001 5mg Every Other Day, Abraxane 60mg/m2 | Phase 1 Level 0 RAD001 5mg Daily, Abraxane 80mg/m2 | Phase 1 Level 1 RAD001 5mg Daily, Abraxane 100mg/m2 | Phase 1 Level 2 RAD001 5mg Daily, Abraxane 125mg/m2 | Phase 1 Level 3 RAD001 10mg Daily, Abraxane 125mg/m2 | Phase II | Total
Number analyzed (Participants) | 0 | 0 | 3 | 6 | 4 | 0 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 1 | 2 | 1 | 0 | 12 | 16
  >=65 years | 0 | 0 | 2 | 4 | 3 | 0 | 2 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 3 | 6 | 4 | 0 | 14 | 27
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 0 | 0 | 3 | 5 | 4 | 0 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 1 | 1 | 0 | 5 | 7
  White | 0 | 0 | 3 | 2 | 3 | 0 | 8 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  |  | 3 | 6 | 4 |  | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Maximum Tolerated Dose (MTD) of RAD001 in Combination of Weekly Abraxane and Determine the Phase II Dose of RAD001.
Time Frame: 5 yrs
Measure: Number; unit: mg
Groups:
- All Participants: Phase I:
  * Abraxane will be given by IV for 30 minutes on the first day of the first three weeks of each 28 day cycle.
  * RAD001 will be given by tablet. The first group of patients will receive RAD001 once daily depending on side effects seen drug could be increased later to twice a day for a 28 day cycle.
  Once a safe and effective drug range is established, the study moves into Phase II.
  Phase II:
  The maximum tolerated dose (established in Phase I) will be given as scheduled below and we will measure the effectiveness of the study drug combination.
  * Abraxane will be given by IV (intravenous infusion) for 30 minutes on the first day of the first three weeks of each 28 day cycle (Day 1, Day 8, and Day 15 of each cycle).
  * RAD001 will be given by tablet based on the dose established in the Phase I part of the study.
  everolimus: Orally administered RAD001 will be initiated at 5 mg daily. Each cohort Phase I: administration will proceed based on escalation criteria. RAD001
Arm/Group | All Participants
Number analyzed (Participants) | 27
mg | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 171 days per patient.
Description: There wer no participants in Level -1, -2 and 3.
Arm/Group | Phase I Level -1 - RAD001 5mg Daily, Abraxane 60mg/m2 | Phase 1 Level -2 - RAD001 5mg Every Other Day, Abraxane 60mg/m2 | Phase 1 Level 0 RAD001 5mg Daily, Abraxane 80mg/m2 | Phase 1 Level 1 RAD001 5mg Daily, Abraxane 100mg/m2 | Phase 1 Level 2 RAD001 5mg Daily, Abraxane 125mg/m2 | Phase 1 Level 3 RAD001 10mg Daily, Abraxane 125mg/m2 | Phase II
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 3/3 | 6/6 | 3/4 | 0/0 | 6/14
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/3 | 2/6 | 0/4 | 0/0 | 4/14
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 2/3 | 6/6 | 4/4 | 0/0 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Level -1 - RAD001 5mg Daily, Abraxane 60mg/m2 (N=0) | Phase 1 Level -2 - RAD001 5mg Every Other Day, Abraxane 60mg/m2 (N=0) | Phase 1 Level 0 RAD001 5mg Daily, Abraxane 80mg/m2 (N=3) | Phase 1 Level 1 RAD001 5mg Daily, Abraxane 100mg/m2 (N=6) | Phase 1 Level 2 RAD001 5mg Daily, Abraxane 125mg/m2 (N=4) | Phase 1 Level 3 RAD001 10mg Daily, Abraxane 125mg/m2 (N=0) | Phase II (N=14)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Alaxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Level -1 - RAD001 5mg Daily, Abraxane 60mg/m2 (N=0) | Phase 1 Level -2 - RAD001 5mg Every Other Day, Abraxane 60mg/m2 (N=0) | Phase 1 Level 0 RAD001 5mg Daily, Abraxane 80mg/m2 (N=3) | Phase 1 Level 1 RAD001 5mg Daily, Abraxane 100mg/m2 (N=6) | Phase 1 Level 2 RAD001 5mg Daily, Abraxane 125mg/m2 (N=4) | Phase 1 Level 3 RAD001 10mg Daily, Abraxane 125mg/m2 (N=0) | Phase II (N=14)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (16)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 7 (19)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (18)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (5)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 10 (16)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 6 (14)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (7)
Dermatology/Skin - (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 12 (43)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Mucositis/stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal - Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bicarbonate, serum-low (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy: sensory (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Mood alteration - Depression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Back (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain - Extremity-limb (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Pain - Head/headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain - Abdomen NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pain - Joint (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Muscle (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain - Dental/teeth/peridontal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Pain NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (7)
Weight loss (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 6 (7)
Edema: head and neck (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (6)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hemorrhage, pulmonary/upper respiratory - Nose (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (4)
Musculoskeletal/Soft Tissue - Othe (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (Infections and infestations) | NA | NA | 1 (1) | 1 (1) | 1 (1) | NA | 0 (0)
Neuropathy (Nervous system disorders) | NA | NA | 1 (1) | 1 (1) | 1 (1) | NA | 0 (0)
hoarseness (Blood and lymphatic system disorders) | NA | NA | 0 (0) | 0 (0) | 1 (1) | NA | 0 (0)
soar throat (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 (0) | 2 (3) | 2 (2) | NA | 0 (0)
Anemia (Blood and lymphatic system disorders) | NA | NA | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | NA | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | NA | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | NA | NA | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT00934895/Prot_SAP_000.pdf